CLINICAL TRIAL: NCT03995420
Title: Virtual Reality Supported Therapy for the Negative Symptoms of Psychosis
Brief Title: VR Therapy for Psychosis Negative Symptoms (V-NeST)
Acronym: V-NeST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Psychiatry, London (Other)
Responsible Party: Principal Investigator, Matteo Cella, Principal Investigator, Institute of Psychiatry, London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 260511
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Psychosis; Schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Virtual Reality Exposure Therapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blind to treatment allocation (single blind)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Therapy (V-NeST) (Experimental): Participants in this arm will receive Virtual Reality Therapy (V-NeST) plus treatment as usual (TAU).
  Interventions: Behavioral: Virtual Reality Therapy (V-NeST); Other: Treatment as Usual
- Treatment as Usual (Other): Participants in this arm will receive treatment as usual (TAU) only.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Virtual Reality Therapy (V-NeST) — V-NeST is a 12-session therapy using psychological intervention principles based on Cognitive Remediation and CBT partly based in Virtual Reality.
  Arms: Virtual Reality Therapy (V-NeST)
Other: Treatment as Usual — multi-modal treatment consisting of different therapies defined by the treating team. These will include regular contact with a care coordinator and medication management by a psychiatrist.

SUMMARY:
Background: Negative symptoms are typically observed in people with schizophrenia and indicate a loss or reduction of a normal function (e.g. reduced motivation and affect display). Despite being important predictors of people's recovery the development of interventions for negative symptoms received only very limited attention. There are currently no evidenced based therapies for these symptoms.

Aims: To test the feasibility and acceptability of a novel virtual reality assisted therapy, called Virtual Reality Supported Therapy for the Negative Symptoms of Psychosis (V-NeST).

Methods: This is a single (rater) blind randomised study with two conditions; V-NeST plus treatment-as-usual (TAU) vs. TAU alone. The study will recruit people with psychosis from NHS community care teams (in England). Assessments will be at baseline and 3-month post-randomisation. A nested qualitative study to identify the key themes associated with the acceptability of the overall study and intervention will be conducted. The study will assess key feasibility parameters such as: consent and availability for screening; eligibility; availability for assessment, randomisation and treatment retention. Acceptability will be assessed by considering: therapy session attendance and drop-out; in-depth feedback from service users interviews; acceptability of the research procedures and measures.

Participants will be assessed with measures of functioning levels and, negative symptoms . Analyses will evaluate the feasibility and analyses of clinical outcomes will be focused on descriptive statistics and confidence intervals for treatment effects. Population variances of the main outcomes will be estimated for future power calculations. A semi-structured interview will explore participants' experience of being recruited to the study, receiving V-NeST and identify barriers (and potential solutions) to treatment engagement.

ELIGIBILITY:
Inclusion Criteria:

* Service users currently under the care of NHS psychosis services;
* Aged over 18;
* in a stable clinical condition (as judged by primary clinician)
* with a documented episode of psychosis and/or a diagnosis of schizophrenia.

Exclusion Criteria:

* Recent antipsychotic medication change (i.e. in the last 3 weeks);
* Moderate to severe learning disability
* Insufficient English for therapy
* Organic impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
the Goal Attainment Scale | 12 weeks
  Measure assessing to degree of participant's individual goals achievement
  Full description of the measure and scoring can be obtained from the reference below:
  Logan TK. Goal Attainment Scaling - Applications, Theory, and Measurement - Kiresuk,Tj, Smith,a, Cardillo,Je. Contemp Psychol. 1995;40(10):984-5.
  Baggio L, Buckley DJ. Detecting change in patient outcomes in a rural ambulatory rehabilitation service: the responsiveness of Goal Attainment Scaling and the Lawton Scale. Aust Health Rev. 2016;40(1):63-8.
  Ng BF, Tsang HW. Evaluation of a Goal Attainment Program using the Goal Attainment Scale for Psychiatric In-patients in vocational rehabilitation. Work. 2000;14(3):209-16.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Psychiatry, King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Still needs to be approved by the sponsor and funder